CLINICAL TRIAL: NCT05939219
Title: Clinical Study on the Consistency of 15-valent Pneumococcal Conjugate Vaccine in Three Batches of 3-month-old Population and the Immunogenicity and Safety of Vaccination in 7-5-year-old Population
Brief Title: Consistency, Immunogenicity, and Safety of Three Batches of 15-valent Pneumococcal Conjugate Vaccine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202204025
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: 15-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 3-month-old group (Experimental): Randomly inoculate 4 batches of 15-valent pneumococcal conjugate vaccine. Immunization program and dosage: Basic immunization at 0, 1, and 2 months, booster immunization at 12-15 months of age, a total of 4 doses administered.
  Dosage form: water injection type
  Interventions: Biological: 15-valent pneumococcal conjugate vaccine 202210001; Biological: 15-valent pneumococcal conjugate vaccineY202210002; Biological: 15-valent pneumococcal conjugate vaccineY202210003; Biological: 15-valent pneumococcal conjugate vaccineY202210004
- 7-11 month old experimental group (Experimental): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: Basic immunization for 0 and 2 months program; Strengthen one dose after 12 months of age; A total of 3 doses were administered.
  Dosage form: water injection type
  Interventions: Biological: 15-valent pneumococcal conjugate vaccineY202210004
- 7-11 month old control group (Active Comparator): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: Basic immunization for 0 and 2 months program; Strengthen one dose after 12 months of age; A total of 3 doses were administered.
  Dosage form: water injection type
  Interventions: Biological: 13 valent pneumococcal polysaccharide conjugate vaccine
- 12-23 months old experimental group (Experimental): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: Immunize 2 doses using the 0 and 2 month program, with a total of 2 doses administered.
  Dosage form: water injection type
  Interventions: Biological: 15-valent pneumococcal conjugate vaccineY202210004
- 12-23 months old control group (Active Comparator): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: Immunize 2 doses using the 0 and 2 month program, with a total of 2 doses administered.
  Dosage form: water injection type
  Interventions: Biological: 13 valent pneumococcal polysaccharide conjugate vaccine
- 2-5 year old experimental group (Experimental): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: 1 dose administered. Dosage form: water injection type
  Interventions: Biological: 15-valent pneumococcal conjugate vaccineY202210004
- 2-5 year old control group (Active Comparator): The experimental group was vaccinated with the 15 valent pneumococcal conjugate vaccine, while the control group was vaccinated with the 13 valent pneumococcal polysaccharide conjugate vaccine, with a ratio of 2:1.
  Immunization program and dosage: 1 dose administered. Dosage form: water injection type
  Interventions: Biological: 13 valent pneumococcal polysaccharide conjugate vaccine

INTERVENTIONS:
Biological: 15-valent pneumococcal conjugate vaccine 202210001 — Immunization program and dosage:3 month old group: basic immunization at 0, 1, and 2 months, and strengthened immunization at 12 to 15 months old, with a total of 4 doses administered. 7-11 month old group: baseline immunization at 0 and 2 months; Strengthen one dose after 12 months of age; A total of 3 doses were administered. 12-23 month old group: Immunized with 2 doses of 0 and 2 month program, a total of 2 doses were administered. 2-5 year old group: 1 dose administered
  Arms: 3-month-old group
Biological: 15-valent pneumococcal conjugate vaccineY202210002 — Immunization program and dosage: 3 month old group: basic immunization at 0, 1, and 2 months, and strengthened immunization at 12 to 15 months old, with a total of 4 doses administered. 7-11 month old group: baseline immunization at 0 and 2 months; Strengthen one dose after 12 months of age; A total of 3 doses were administered. 12-23 month old group: Immunized with 2 doses of 0 and 2 month program, a total of 2 doses were administered. 2-5 year old group: 1 dose administered
  Arms: 3-month-old group
Biological: 15-valent pneumococcal conjugate vaccineY202210003 — Immunization program and dosage: 3 month old group: basic immunization at 0, 1, and 2 months, and strengthened immunization at 12 to 15 months old, with a total of 4 doses administered. 7-11 month old group: baseline immunization at 0 and 2 months; Strengthen one dose after 12 months of age; A total of 3 doses were administered. 12-23 month old group: Immunized with 2 doses of 0 and 2 month program, a total of 2 doses were administered. 2-5 year old group: 1 dose administered
  Arms: 3-month-old group
Biological: 15-valent pneumococcal conjugate vaccineY202210004 — Immunization program and dosage: 3 month old group: basic immunization at 0, 1, and 2 months, and strengthened immunization at 12 to 15 months old, with a total of 4 doses administered. 7-11 month old group: baseline immunization at 0 and 2 months; Strengthen one dose after 12 months of age; A total of 3 doses were administered. 12-23 month old group: Immunized with 2 doses of 0 and 2 month program, a total of 2 doses were administered. 2-5 year old group: 1 dose administered
  Arms: 12-23 months old experimental group; 2-5 year old experimental group; 3-month-old group; 7-11 month old experimental group
Biological: 13 valent pneumococcal polysaccharide conjugate vaccine — Immunization program and dosage: 7-11 month old group: baseline immunization at 0 and 2 months; Strengthen one dose after 12 months of age; A total of 3 doses were administered. 12-23 month old group: Immunized with 2 doses of 0 and 2 month program, a total of 2 doses were administered. 2-5 year old group: 1 dose administered
  Arms: 12-23 months old control group; 2-5 year old control group; 7-11 month old control group

SUMMARY:
The objective of this clinical trial is to evaluate the consistency of the 15-valent pneumococcal conjugate vaccine in three batches of the 3-month-old population, as well as the immunogenicity and safety of vaccination in the 7-5-year-old population

DETAILED DESCRIPTION:
The purpose of this experiment

1. evaluate the consistency of clinical immune efficacy of three batches of commercially produced 15-valent pneumococcal conjugate vaccines.
2. Compare the immunogenicity of commercial scale produced 15-valent pneumococcal conjugate vaccines in the 3-month-old population with the immunogenicity (non inferiority) of pilot scale produced 15-valent pneumococcal conjugate vaccines, that is, a clinical bridging study between commercial scale vaccines and Phase III clinical trial vaccines.
3. Evaluate the immunogenicity and safety of the 15-valent pneumococcal conjugate vaccine in the 7-5-year-old population after vaccination.

The commercial three batches and pilot scale batches were designed using a randomized, double-blind, parallel controlled trial of different batches of vaccines. The commercial three batches adopt equivalence design, and the immunogenicity results of the three batches are merged on the basis of equivalence, and compared with the immunogenicity of the pilot scale batch for non-inferiority.

Compare the immunogenicity data of the 7-5-year-old population experimental group with the immunogenicity results of the 3-month-old group (after merging three commercial batches on an equivalent basis) at the basic immune stage for non-inferiority.

At the same time, a positive control was established in the 7-month-5-year-old population, and a randomized, blind design was used to compare the immunogenicity of the experimental group and the control group in this age group.

The study population consists of a total of 2346 people, including 1104 people at the age of 3 months, divided into four groups with 276 people in each group. They were assigned to batch 1, batch 2, batch 3, and the pilot scale module at a ratio of 1:1:1:1. There are a total of 1242 people aged 7 months to 5 years old, divided into three age groups: 7-11 months old, 12-23 months old, and 2-5 years old, with 414 people in each age group. Three age groups of participants were randomly assigned to the experimental group or control group in a 2:1 ratio. The experimental group received a 15-valent pneumococcal conjugate vaccine (batch 3), while the control group received a 13-valent pneumococcal polysaccharide conjugate vaccine produced by Yuxi Watson Biotechnology Co., Ltd. Among them:

1. 3 months old: Basic immunization according to the 0, 1, and 2 month program (window period:+10 days); Strengthen immunization with 1 dose at the age of 12-15 months.
2. 7-11 months of age: basic immunization with a 0 to 2-month program (window period:+10 days); After 12 months of age, strengthen the vaccination with 1 dose (3rd dose), with a minimum interval of 2 months between the 2nd dose.
3. 12-23 months old: Immunize with 2 doses of 0 and 2 month program. The interval between two doses of vaccination should be at least 2 months (window period:+10 days).
4. 2-5 years old: receive 1 dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants and children aged 3 months, 7 months, and 5 years old;
* Infants under 1 year old should be born at full term (37 to 42 weeks of pregnancy) and have a birth weight within the range of (2500g ≤ body weight ≤ 4500g);
* After informed consent, the Legal guardian voluntarily signs the informed consent form and can comply with the requirements of the clinical research scheme;
* The subject has no history of receiving other live attenuated vaccines within ≤ 14 days, and no history of receiving other non live vaccines within ≤ 7 days;
* Underarm temperature ≤ 37.0 ℃.

Exclusion Criteria:

* Previously received commercially available or experimental pneumococcal vaccines;
* Have a history of invasive disease caused by Streptococcus pneumoniae that has been confirmed by culture in the past;
* Have a history of severe allergies to vaccines or medication;
* Have a history of Nervous system disease such as convulsion, epilepsy, nervous system tumor, craniocerebral trauma, psychiatric history or family history;
* Babies born under the age of 1 year with severe abnormal birth process (such as instrumental delivery) or a history of asphyxia or neurological organ damage;
* Patients with pathological jaundice confirmed by current diagnosis;
* A history of clearly diagnosed thrombocytopenia or other coagulation disorders may lead to contraindications for injection;
* Immunoglobulin or any blood products (except hepatitis B immunoglobulin) were given within 3 months before enrollment;
* Known or suspected to have immunological function defects, and received long-term Immunosuppressive drug treatment (radiotherapy, chemotherapy, Corticosteroid, antimetabolics, cytotoxic drugs), HIV infection or HIV infected parents within six months before vaccination;
* Having severe congenital malformations, severe malnutrition, developmental disorders, or genetic defects (such as broad bean disease);
* Currently suffering from serious chronic disease, infectious disease, active infection, liver disease, kidney disease, cardiovascular disease, and malignant tumor;
* Absence of spleen or deficiency of spleen function caused by any circumstances;
* Systemic rash, skin ringworm, skin suppuration or blisters;
* Participating in other clinical trials;
* Any situation that the researcher believes may affect the evaluation of the study.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2346 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean concentration of vaccine Serotype specific pneumococcal IgG antibody | 30 days after basic immunization at 3 months old and 7-11 months old, and 30 days after full immunization at 12-23 months old and 2-5 years old
  Immunogenicity evaluation
Vaccine Serotype specific pneumococcal IgG antibody concentration ≥ 0.35 μg/ml of proportion of subjects | 30 days after basic immunization at 3 months old and 7-11 months old, and 30 days after full immunization at 12-23 months old and 2-5 years old
  Immunogenicity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Hebei Provincial Center for Disease Control and Prevention, Shijiangzhuang, Hebei, China